CLINICAL TRIAL: NCT05602077
Title: The Diagnostic Accuracy of Sonography in Indirect Elbow Trauma Compared With Plain X-ray: a Prospective Single Centre Comparative Diagnostic Accuracy Study
Brief Title: Accuracy of Sonography in Elbow Trauma
Acronym: SONOELB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eckehart SCHÖLL (Other)
Collaborators: Basel Academy for Quality and Research in Medicine; Prof. Dr. Werner Vach (Statistician) (Unknown); Merian Iselin Klinik; Anja Mair (medical specialist) (Unknown); Merian Iselin Klinik; Dr. Thomas Egelhof (head of radiology) (Unknown)
Responsible Party: Sponsor-Investigator, Eckehart SCHÖLL, Head of Emergency Department, Merian Iselin Klinik
Organization: Merian Iselin Klinik (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SONOELB_Vs_2022_09_12_1.1
Record Dates: First submitted 2022-10-22; First posted 2022-11-01 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Elbow Fracture; Radial Head Fracture; Elbow Sprain; Coronoid Process Fracture; Distal Humerus Fracture
Keywords: elbow; ultrasound; radial head
MeSH Terms: conditions — Elbow Fractures; Radial Head and Neck Fractures; Humeral Fractures, Distal

STUDY DESIGN:
Intervention Model Description: Prospective single centre comparative diagnostic accuracy study
Masking Description: The two modalities to be compared (POCUS and XR) and the reference standard (CBCT) will be applied in a consecutive series of 130 patients with a suspicion of an indirect elbow fracture at the emergency department of a single center. All investigations will be part of the initial, single visit of the patient at the emergency department.
  The modalities will be evaluated blinded for each other. The design is well known as a comparative, paired accuracy study. The design allows to estimate the accuracy of the two diagnostic modalities and the corresponding difference as well as the agreement between the two modalities.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- POCUS and Control Intervention (Experimental): POCUS: Point of care ultrasound
  Control-Intervention: X-ray examination and Cone Beam Computed Tomography (CBCT)
  Interventions: Device: POCUS

INTERVENTIONS:
Device: POCUS — POCUS: The ultrasound examination of the injured elbow includes seven standard settings. The probe is placed on the joint in four ventral and in three posterior positions. If hemarthrosis is detected, this is always suspicious of a possible intra-articular fracture. Even the smallest amounts of blood can be detected sonographically. The surfaces of the bones involved in the joint (humerus, ulna, radius) are accurately displayed in all seven sonography settings. Disrupted bone surface indicates a fracture.
  XR: The conventional radiograph of the injured elbow consists of three standard views: ap, lateral and Norman oblique.
  CBCT: The injured elbow is placed in an almost most extended position in the CBCT tube.
  Other Names: Control Intervention: XR / CBCT

SUMMARY:
X-rays (XR) are today the standard modality for the diagnosis of bone fractures in the lower or upper limbs in the emergency room. Point-of-care ultrasound (POCUS) is an alternative with some obvious advantages especially in the emergency room setting: It does not require the patient to fix the bone of interest in a stable position, allows observing the bone and joints under movement by the patient, can be performed at bedside, and avoids the exposure to radiation.

The advances in ultrasound technology has increased the interest in using POCUS as an alternative to XR in recent years. POCUS is used routinely prior to XR at the ORTHO-NOTFALL of the Merian Iselin Klinik Basel (MIK) in patients with suspicion for an indirect elbow trauma. It is the aim of this project to use this constellation in order to contribute to a systematic comparison of the value of the two modalities with the long-term aim to establish POCUS as the first-line diagnostic tool.

As a fist project, the SONOELB study was initiated. This study aims at a comparison of the diagnostic accuracy between XR and POCUS using CT as reference. The project started in October 2022 and aims at enrolling 130 patients until March 2025. The project is financially supported by the Merian Iselin Science Research PLC.

DETAILED DESCRIPTION:
Objective:

The primary objective is to compare the diagnostic accuracy of POCUS and XR with respect to diagnosing fractures of the elbow after an indirect elbow trauma in the ED setting and to investigate the rate of agreement between the two modalities.

The primary outcome is the difference in diagnostic accuracy between the two modalities with respect to diagnosing a radial head fracture and the degree of agreement between the two modalities.

Secondary outcomes are the difference in diagnostic accuracy between the two modalities and the rate of agreement with respect to the other fracture types, to the decisions "any fracture", and to the decision "any fracture other than radial head".

Experimental Intervention (medical device) POCUS: The ultrasound examination of the injured elbow includes seven standard settings. The probe is placed on the joint in four ventral and in three posterior positions. If hemarthrosis is detected, this is always suspicious of a possible intra-articular fracture. Even the smallest amounts of blood can be detected sonographically.

The surfaces of the bones involved in the joint (humerus, ulna, radius) are accurately displayed in all seven sonography settings. Disrupted bone surface indicates a fracture.

POCUS will be performed according to the local SOP.

Control Intervention (standard/routine/comparator) XR: The conventional radiograph of the injured elbow consists of three standard views: ap, lateral and Norman oblique. This X-ray examination is the most commonly performed technique to date to diagnose an injured elbow.

CBCT (Cone Beam Computed Tomography): The injured elbow is placed in an almost most extended position in the CBCT tube. For this purpose, the affected arm is placed and fixed on a carbon-splint. The examination time is about 40 seconds XR will be performed according to the standard procedures of the ED of the MIK. The same holds for CBCT.

Any of the three diagnostic procedures applied can be discontinued in the case of patient discomfort, harm, or risk of harm according to the standard procedures of the MIK.

Compliance of the staff of the ED with performing the three modalities is supported by SOPs and internal training.

In the case of withdrawal of a patient, the reasons are recorded on the CRF. The data of these patients will not be included in the statistical analysis. The data will not be deleted in the data management system. Patients who withdraw themselves are offered a chat with the PI and further consultations.

Patients included in the trial will follow the standard management at the MIK. There are only two changes:

* a CBCT is performed in addition after having performed both POCUS and XR, if there are no positive findings on POCUS or XR.
* an additional blinded evaluation of all CBCTs will be done by one independent rater.

CBCT will be ordered by the staff of the ED in all patients and may be preliminary evaluated. However, these evaluations will not be documented as part of this study. They are also not accessible for the staff at the Radiology Department in the routine evaluation of the XRs.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent signed by the subject
* Suspicion for an indirect elbow trauma as part of the routine management at the ED of the MIK.

Exclusion Criteria:

* Age below 18
* Patients who are lacking capacity of judgment
* Patients with (temporary) cognitive impairment which makes an understanding of the patient information unlikely
* Patients with limited knowledge of German or English which makes an understanding of the patient information unlikely
* Patients with contraindications for US, XR or CT.
* Lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Difference in diagnostic accuracy of sonography in radial head fractures compared with plain x-ray | within the emergency department stay (1 day)
  In order to assess the diagnostic accuracy, CBCT is used as a reference standard in all patients.
  The findings from the POCUS, XR, and CBCT with respect to a fracture of the radial head are documented on three different CRFs: POCUS, XR, CBCT.
  CRF POCUS (7 views): unaffected(Y/N) - haemarthros (y/n) - fractures of the different parts CRF XR: (ap/lateral/Norman): unaffected(Y/N) - fat pad sign (y/n) - fractures of the different parts CRF CBCT: unaffected(Y/N) - fractures of the different parts

SECONDARY OUTCOMES:
Difference in diagnostic accuracy of sonography in other elbow fractures compared with plain x-ray: Fossa olecrani | within the emergency department stay (1 day)
  difference in diagnostic accuracy between the two modalities and the rate of agreement with respect to the other fracture types, to the decisions "any fracture", and to the decision "any fracture other than radial head".
  Fossa olecrani fractures as part of the distal humerus
  CRF POCUS (7 views): unaffected(Y/N) - haemarthros (y/n) - fractures of the different parts CRF XR: (ap/lateral/Norman): unaffected(Y/N) - fat pad sign (y/n) - fractures of the different parts CRF CBCT: unaffected(Y/N) - fractures of the different parts
Difference in diagnostic accuracy of sonography in other elbow fractures compared with plain x-ray: supracondylar fracture | within the emergency department stay (1 day)
  difference in diagnostic accuracy between the two modalities and the rate of agreement with respect to the other fracture types, to the decisions "any fracture", and to the decision "any fracture other than radial head".
  Supracondylar fractures as part of the distal humerus
  CRF POCUS (7 views): unaffected(Y/N) - haemarthros (y/n) - fractures of the different parts CRF XR: (ap/lateral/Norman): unaffected(Y/N) - fat pad sign (y/n) - fractures of the different parts CRF CBCT: unaffected(Y/N) - fractures of the different parts
Difference in diagnostic accuracy of sonography in other elbow fractures compared with plain x-ray: condylar fracture | within the emergency department stay (1 day)
  difference in diagnostic accuracy between the two modalities and the rate of agreement with respect to the other fracture types, to the decisions "any fracture", and to the decision "any fracture other than radial head".
  medial or lateral fractures as part of the distal humerus
  CRF POCUS (7 views): unaffected(Y/N) - haemarthros (y/n) - fractures of the different parts CRF XR: (ap/lateral/Norman): unaffected(Y/N) - fat pad sign (y/n) - fractures of the different parts CRF CBCT: unaffected(Y/N) - fractures of the different parts
Difference in diagnostic accuracy of sonography in other elbow fractures compared with plain x-ray: capitulum humeri fracture | within the emergency department stay (1 day)
  difference in diagnostic accuracy between the two modalities and the rate of agreement with respect to the other fracture types, to the decisions "any fracture", and to the decision "any fracture other than radial head".
  capitulum humeri fracture as part of the distal humerus
  CRF POCUS (7 views): unaffected(Y/N) - haemarthros (y/n) - fractures of the different parts CRF XR: (ap/lateral/Norman): unaffected(Y/N) - fat pad sign (y/n) - fractures of the different parts CRF CBCT: unaffected(Y/N) - fractures of the different parts
Difference in diagnostic accuracy of sonography in other elbow fractures compared with plain x-ray: Coronoid process fracture | within the emergency department stay (1 day)
  difference in diagnostic accuracy between the two modalities and the rate of agreement with respect to the other fracture types, to the decisions "any fracture", and to the decision "any fracture other than radial head".
  Coronoid process fracture as part of the proximal ulna
  CRF POCUS (7 views): unaffected(Y/N) - haemarthros (y/n) - fractures of the different parts CRF XR: (ap/lateral/Norman): unaffected(Y/N) - fat pad sign (y/n) - fractures of the different parts CRF CBCT: unaffected(Y/N) - fractures of the different parts
Difference in diagnostic accuracy of sonography in other elbow fractures compared with plain x-ray: Olecranon fracture | within the emergency department stay (1 day)
  difference in diagnostic accuracy between the two modalities and the rate of agreement with respect to the other fracture types, to the decisions "any fracture", and to the decision "any fracture other than radial head".
  Olecranon fracture as part of the proximal ulna
  CRF POCUS (7 views): unaffected(Y/N) - haemarthros (y/n) - fractures of the different parts CRF XR: (ap/lateral/Norman): unaffected(Y/N) - fat pad sign (y/n) - fractures of the different parts CRF CBCT: unaffected(Y/N) - fractures of the different parts

CONTACTS AND LOCATIONS:
Locations (1):
- Merian Iselin Klinik, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tsou PY, Ma YK, Wang YH, Gillon JT, Rafael J, Deanehan JK. Diagnostic accuracy of ultrasound for upper extremity fractures in children: A systematic review and meta-analysis. Am J Emerg Med. 2021 Jun;44:383-394. doi: 10.1016/j.ajem.2020.04.071. Epub 2020 Apr 27. PMID 32507477
- [Result] Pourmand A, Shokoohi H, Maracheril R. Diagnostic accuracy of point-of-care ultrasound in detecting upper and lower extremity fractures: An evidence-based approach. Am J Emerg Med. 2018 Jan;36(1):134-136. doi: 10.1016/j.ajem.2017.06.052. Epub 2017 Jun 27. No abstract available. PMID 28669695
- [Result] Champagne N, Eadie L, Regan L, Wilson P. The effectiveness of ultrasound in the detection of fractures in adults with suspected upper or lower limb injury: a systematic review and subgroup meta-analysis. BMC Emerg Med. 2019 Jan 28;19(1):17. doi: 10.1186/s12873-019-0226-5. PMID 30691395
- [Result] Hanlon DP, Mavrophilipos V. The Emergent Evaluation and Treatment of Elbow and Forearm Injuries. Emerg Med Clin North Am. 2020 Feb;38(1):81-102. doi: 10.1016/j.emc.2019.09.005. PMID 31757256
- [Result] Bianchi S. Ultrasound and bone: a pictorial review. J Ultrasound. 2020 Sep;23(3):227-257. doi: 10.1007/s40477-020-00477-4. Epub 2020 May 17. PMID 32419074
- [Result] De Maeseneer M, Jacobson JA, Jaovisidha S, Lenchik L, Ryu KN, Trudell DR, Resnick D. Elbow effusions: distribution of joint fluid with flexion and extension and imaging implications. Invest Radiol. 1998 Feb;33(2):117-25. doi: 10.1097/00004424-199802000-00010. PMID 9493728
- [Result] Rutten MJ, Collins JM, de Waal Malefijt MC, Kiemeney LA, Jager GJ. Unsuspected sonographic findings in patients with posttraumatic shoulder complaints. J Clin Ultrasound. 2010 Nov-Dec;38(9):457-65. doi: 10.1002/jcu.20745. PMID 20848574
- [Result] Malahias MA, Manolopoulos PP, Kadu V, Shahpari O, Fagkrezos D, Kaseta MK. Bedside Ultrasonography for Early Diagnosis of Occult Radial Head Fractures in Emergency Room: A CT-Comparative Diagnostic Study. Arch Bone Jt Surg. 2018 Nov;6(6):539-546. PMID 30637310
- [Result] Avci M, Kozaci N, Beydilli I, Yilmaz F, Eden AO, Turhan S. The comparison of bedside point-of-care ultrasound and computed tomography in elbow injuries. Am J Emerg Med. 2016 Nov;34(11):2186-2190. doi: 10.1016/j.ajem.2016.08.054. Epub 2016 Aug 27. PMID 27645809
- [Result] Waterbrook AL, Adhikari S, Stolz U, Adrion C. The accuracy of point-of-care ultrasound to diagnose long bone fractures in the ED. Am J Emerg Med. 2013 Sep;31(9):1352-6. doi: 10.1016/j.ajem.2013.06.006. Epub 2013 Jul 26. PMID 23891601
- [Result] Avci M, Kozaci N, Tulubas G, Caliskan G, Yuksel A, Karaca A, Doganay F, Etli I. Comparison of Point-of-Care Ultrasonography and Radiography in the Diagnosis of Long-Bone Fractures. Medicina (Kaunas). 2019 Jul 9;55(7):355. doi: 10.3390/medicina55070355. PMID 31324028
- [Result] Eckert M, Vach W. On the use of comparison regions in visualizing stochastic uncertainty in some two-parameter estimation problems. Biom J. 2020 May;62(3):598-609. doi: 10.1002/bimj.201800232. Epub 2019 Oct 29. PMID 31661558